CLINICAL TRIAL: NCT05519462
Title: Low-Dose CBCT Protocol for Pre-Surgical Evaluation of the Mandibular Third Molar, a Feasible Choice?
Status: Completed | Type: Observational
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Kristina Hellén-Halme, Professor, Malmö University
Other Study IDs: FO2020-242
Record Dates: First submitted 2022-08-24; First posted 2022-08-29 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Teeth; Lesion; Tooth Diseases
Keywords: CBCT
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Low-Dose CBCT Protocol for Pre-Surgical Evaluation of the Mandibular Third Molar.

CBCT investigations with standard and low dose protocol for evalutation of the mandibular third molar.

DETAILED DESCRIPTION:
Two CBCT scans were acquired of each examination site: one scan using the standard clinical protocol (90kV, 5mA, 9.4s) and one, the low-dose protocol (90kV, 2mA, 9.4s). All exposures were made with a Veraviewepocs 3D F40 (J Morita Corp.; Kyoto, Japan) using a field of view (FOV) of 4.0 x 4.0 cm and a rotation mode of 180°, voxel size of 0.125 mm.

ELIGIBILITY:
Inclusion Criteria:

* a need for a CBCT investigation of the mandibula third molar

Exclusion Criteria:

* been involved in radiographic examinations for science beforer.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adults
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
evaluation of radiographic images | 1 day
  landmarks

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Hellen-Halme, professor, Study Chair — Malmö University
Locations (1):
- Kristina Hellen-Halme, Malmo, Sweden